CLINICAL TRIAL: NCT01128465
Title: Investigation on the Pharmacokinetic and -Dynamic of Propofol During Awake Craniotomy
Brief Title: Pharmacokinetic and -Dynamic of Propofol During Awake Craniotomy
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Martin Soehle, MD, DESA, Dept. of Anaesthesiology and Intensive Care Medicine
Other Study IDs: AC
Record Dates: First submitted 2010-02-22; First posted 2010-05-24 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Brain Tumor
Keywords: propofol; awake craniotomy; patients requiring an awake craniotomy for brain tumor/lesion resection
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Certain kind of neurosurgical procedures require intraoperative alertness of the patient, for example to perform speech tests during brain tumor resection. With respect to anaesthesia, it is therefore required that the patient is asleep during the beginning and the end of the procedure, however fully awake in between. To do so, the anaesthetic propofol is used and an accurate knowledge of its pharmacokinetic and -dynamic (pk/pd) parameters is required to optimally control anaesthesia. However, diverse pk/pd-parameter sets have been described in the literature.

The aim of the study is to investigate whether the pk/pd model proposed by Marsh et al. or by Schnider et al. more accurately describe the pk/pd of propofol during awake craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for awake craniotomy

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a University Hospital requiring an awake craniotomy for resection of a brain tumor or lesion
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
prediction error for propofol plasma concentrations | day of surgery (day 1)
  On the day of surgery, plasma samples will be drawn during induction, maintenance and recovery from anesthesia. Subsequently the actually measured propofol plasma concentration will be compared with the predicted propofol plasma concentration (according to Marsh et al. and Schnider et al.), and the prediction error will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Soehle, MD, DESA, D habil, Principal Investigator — Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Germany
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, Univ. of Bonn, Bonn, Germany

REFERENCES:
- [Background] Schnider TW, Minto CF, Gambus PL, Andresen C, Goodale DB, Shafer SL, Youngs EJ. The influence of method of administration and covariates on the pharmacokinetics of propofol in adult volunteers. Anesthesiology. 1998 May;88(5):1170-82. doi: 10.1097/00000542-199805000-00006. PMID 9605675
- [Background] Marsh B, White M, Morton N, Kenny GN. Pharmacokinetic model driven infusion of propofol in children. Br J Anaesth. 1991 Jul;67(1):41-8. doi: 10.1093/bja/67.1.41. PMID 1859758
- [Derived] Soehle M, Wolf CF, Priston MJ, Neuloh G, Bien CG, Hoeft A, Ellerkmann RK. Comparison of propofol pharmacokinetic and pharmacodynamic models for awake craniotomy: A prospective observational study. Eur J Anaesthesiol. 2015 Aug;32(8):527-34. doi: 10.1097/EJA.0000000000000255. PMID 25774459